CLINICAL TRIAL: NCT05692505
Title: Multicenter Performance Study of QuadQuik Invitro Diagnostic Device
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Genlantis Diagnostics (Industry)
Collaborators: Ahsan Awan (Unknown)
Responsible Party: Sponsor
Other Study IDs: genl-qq-1
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections; Hepatitis C; Hepatitis B; Syphilis Infection
MeSH Terms: conditions — HIV Infections; Hepatitis C; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Positive test subjects: Subjects having previous positive tests verified by certified laboratory
  Interventions: Diagnostic Test: QuadQuik
- Control subjects: Subjects having no previous positive tests verified by certified laboratory
  Interventions: Diagnostic Test: QuadQuik

INTERVENTIONS:
Diagnostic Test: QuadQuik — Invitro diagnostic device

SUMMARY:
To Demonstrate Clinical Performance of the TriQuik Invitro Diagnostic Device

DETAILED DESCRIPTION:
Measurement Methodology Whole blood samples are collected by fingerstick. Samples tested immediately.

Using the supplied sample dropper, transfer specimen blood drop into the two sample wells. Wait 20-30 seconds. Add two drops of the supplied assay buffer (~90µL) to the same sample wells Read result in 20 mins.

Primary end points will determine how accurate these tests are (p<=0.02) by analyzing for:

Diagnostic Sensitivity; TP / (TP + FN) The ability of the test to correctly identify those patients with the disease Diagnostic Specificity; TN / (TN + FP) The ability of the test to correctly identify those patients who are truly free of the specific disease Positive Predictive Value: TP / (TP+ FP) The probability that subjects with a positive test truly have the disease. Negative Predictive Value: TN / (FN + TN) The probability that subjects with a negative test truly don't have the disease.

An estimated 200 patients are to be enrolled as follows:

150 with a documented medical history of HIV, HBV, HCV or Syphilis. A combination of 2 or 3 conditions is acceptable.

HbsAg patients need to have a HbsAg on file < 2 years. HIV and HCV or Syphilis patients only need one antibody test in their medical chart.

50 with no documented medical history of HIV, HBV, HCV or Syphilis and are considered normal.

Male or female subjects, ages ≥18 years.

ELIGIBILITY:
Inclusion Criteria:

a documented medical history of HIV, HBV, HCV or syphilis. A combination of 2 or 3 conditions is acceptable.

HbsAg patients need to have a HbsAg on file < 2 years. HIV and HCV patients only need one antibody test in their medical chart. no documented medical history of HIV, HBV, HCV or syphilis and are considered normal.

Male or female subjects, ages ≥18 years. Signed informed consent provided by an authorized subject representative (based on local Institutional Review Board (IRB)/ethics panel requirements).-

Exclusion Criteria:

Any other condition or prior therapy, which, in the opinion of the investigator, would make the subject unsuitable for this study.

Participation in any phase of another clinical research study involving the evaluation of another investigational drug or device within 30 days before randomization.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study patients are seen, recruited and consented from local clinics and physician offices.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Standard performance criteria | <1 day
  Diagnostic Sensitivity, Diagnostic Specificity, Positive Predictive Value, Negative Predictive Value

CONTACTS AND LOCATIONS:
Locations (1):
- Genlantis Diagnostics, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided